CLINICAL TRIAL: NCT06919510
Title: A Phase ll Study of Neoadjuvant Short-course Radiotherapy Followed by Lvonescimab and Chemotherapy Versus Neoadjuvant Short-course Radiotherapy Followed by Chemotherapy in pMMR/MSS Locally Advanced Rectal Cancer
Brief Title: A Phase ll Study of Neoadjuvant Short-course Radiotherapy Followed by Ivonescimab and Chemotherapy in pMMR/MSS Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Akeso (Industry)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, President, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-016
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Short-course radiotherapy followed by ivonescimab and chemotherapy) (Experimental): Subjects will receive short-course radiotherapy of 25Gy/5 fractions, followed by neoadjuvant chemotherapy of CAPOX and ivonescimab. After neoadjuvant treatment, the patients and investigator could choose one of the following treatments:(1) Surgery. The patients will receive surgery within 4-8 weeks after the last dose of capecitabine, and the surgical method is selected by the investigator: (2) Watch and Wait(only for patients with clinical complete response after neoadjuvant therapy).
  Interventions: Drug: lvonescimab; Drug: CAPOX (oxaliplatin/capecitabine); Radiation: radiotherapy; Procedure: Surgery or watch&wait
- Group B (Short-course radiotherapy followed by chemotherapy) (Active Comparator): Subjects will receive short-course radiotherapy of 25Gy/5 Fraction, followed by neoadjuvant chemotherapy of CAPOX .After neoadiuvant treatment, the patients and investigator could choose one of the following treatments:(1) Surgery. The patients will receive surgery within 4-8 weeks after the last dose of capecitabine, and the surgical method is selected by the investigator; (2) Watch and Wait (only for patients with clinical complete response after neoadjuvant therapy).
  Interventions: Drug: CAPOX (oxaliplatin/capecitabine); Radiation: radiotherapy; Procedure: Surgery or watch&wait

INTERVENTIONS:
Drug: lvonescimab — lvonescimab, DS1, D1,q3w, intravenous infusion
  Arms: Group A (Short-course radiotherapy followed by ivonescimab and chemotherapy)
Drug: CAPOX (oxaliplatin/capecitabine) — Oxaliplatin 130 mg / m2, D1, intravenous infusion, q3w, Capecitabine 1000 mg / m2,twice a day, oral,1-14 days, then rest for 7 days, q3w.
Radiation: radiotherapy — 5* 5Gy, once a day, 5Gy each time, for 5 days
Procedure: Surgery or watch&wait — The surgical method is selected by the investigator. Watch and Wait (only for patients with clinical complete response after neoadjuvant therapy)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of short-course radiotherapy followed by ivonescimab and chemotherapy in participants with pMMR/MSS locally advanced rectal cancer. Patients were randomly assigned to experimental group A or control group B according to a 1:1 ratio. In group A, patients will receive neoadjuvant short-course radiotherapy followed by ivonescimab and chemotherapy. In group B, patients will receive neoadjuvant short-course radiotherapy followed by chemotherapy. After neoadjuvant treatment, the patients and investigator could choose one of the following treatments:(1) Surgery. The patients will receive surgery within 4-8 weeks after the last dose of capecitabine, and the surgical method is selected by the investigator, (2) Watch and Wait (only for patients with clinical complete response after neoadjuvant therapy).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years;
2. ECOG perfommance status of 0 or 1;
3. Life expectancy: more than 2 years;
4. Histologically proven rectal adenocarcinoma;
5. Tumor biopsy immunohistochemistry proven pMMR, positive for four proteins, MLH1, MSH2, MSH6 and PMS2, or MSS determined by gene testing;
6. According to the 8th Edition of the AJCC Staging Manual, clinical stage cT3-4NanyM0 or cTxN+M0 of II-III rectal cancer was determined by Magnetic resonance imaging (MRI)±transrectal ultrasonography/ ultrasound endoscopy. Lower edge of the tumor was ≤ 12 cm from the anal verge;
7. Eligible for R0 surgery;
8. No prior anti-tumor treatment for rectal cancer,including radiotherapy,chemotherapy, immunotherapy, biologics, small molecule targeted therapy, etc;
9. Adequate organ function;
10. Males or females with reproductive ability who are willing to use contraception in the trial;

Exclusion Criteria:

1. Any distant metastasis or inoperable disease, regardless clinical stage;
2. Previous (within 5 years) or concurrent other malignant tumors, excluding those that have been cured;
3. Current presence of gastric intestine obstruction, bleeding or perforation which need emergency surgery;
4. Multiple primary rectal cancers;
5. Previous pelvic or abdominal radiotherapy;
6. Difficulty swallowing;
7. Current presence of uncontrolled combined disease;
8. Active clinical infections;
9. History of severe bleeding tendency or coagulation dysfunction;
10. Presence or history of immunodeficiency; positive for HIV antibodies, current long-term use of systemic corticosteroids or other immunosuppressants;
11. Subjects with known active tuberculosis (TB); suspected active TB should be excluded by clinical examination, known active syphilis infection;
12. Received a live vaccine within 30 days prior to the study, or plan to receive a live vaccine during the study;
13. Local or systemic disease caused by non-malignancy, or disease or symptom secondary to tumor, that can lead to higher medical risk and/or uncertainty in survival;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through study completion, an average of 6 month
  Adverse events and surgical safety
Complete response rate | 4 weeks after curative surgery for pCR; 2-4 weeks after the completion of neoadjuvant therapy (last dose of capecitabine) for cCR
  The proportion of CR cases (pCR for those who underwent surgery and cCR for those who didn't receive surgery)
Clinical complete response rate | 2-4 weeks after the completion of neoadjuvant therapy (last dose of capecitabine)
  The proportion of clinical complete response cases.

SECONDARY OUTCOMES:
Pathologic complete response | 4 weeks after surgery
  The proportion of pathologic complete response cases for those who underwent surgery
TRG | 4 weeks after surgery
  Tumor regression grade according to AJCC TRG grading system
R0 resection rate | 4 weeks after surgery
  R0 resection rate
Local recurrence | 3 years after Randomization
  Local recurrence
Distant metastasis | 3 years after Randomization
  Distant metastasis
OS | 3 years after Randomization
  Overall survial
EFS | 3 years after Randomization
  Event free of survival

IPD SHARING:
Plan to Share IPD: Undecided